CLINICAL TRIAL: NCT06624319
Title: Comparing the Analgesic Effect of Two Different Doses of Dexmedetomidine Added to Bupivacaine in Ultrasound-guided Transversus Abdominis Plane Block in Patients Undergoing Lower Abdominal Cancer Surgeries; A Randomized Clinical Trial
Brief Title: Two Doses of Dexmedetomidine as Adjuvent to Bupivacaine in Tap Block
Acronym: Dexmed/tap
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Salama Tawfeek, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2024-200895
Record Dates: First submitted 2024-09-28; First posted 2024-10-02 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Pain
Keywords: Tap block; Dexmedetomidine
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients will receive pre-emptive ultrasound-guided tap block with two different doses of dexmedetomidine in 20 ml volume added to 20 mL of 0.25% bupivacaine (40 ml in total) 20 ml will be applied on each side of the abdominal wall after induction of GA.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tap block with 0.5 μg/kg dexmedetomidine (Active Comparator): will receive pre-emptive ultrasound-guided tap block with 0.5 μg/kg dexmedetomidine in 20 ml volume added to 20 mL of 0.25% bupivacaine (40 ml in total) 20 ml will be applied on each side of the abdominal wall after induction of GA.
  Interventions: Drug: Dexmedetomidine as adjuvent to bupvacaine in tap block
- tap block with 1.5 μg/kg dexmedetomidine (Active Comparator): will receive pre-emptive ultrasound-guided tap block with 1.5 μg/kg dexmedetomidine in 20 ml volume added to 20 mL of 0.25% bupivacaine (40 ml in total) 20 ml will be applied on each side of the abdominal wall after induction of GA.
  Interventions: Drug: Dexmedetomidine as adjuvent to bupvacaine in tap block

INTERVENTIONS:
Drug: Dexmedetomidine as adjuvent to bupvacaine in tap block — The analgesic effect of Two different doses of dexmedetomidine as adjuvent to bupivacaine in tap block
  Other Names: Precedex

SUMMARY:
The aim of this study to determine the optimal dose of dexmedetomidine as an adjuvant to bupivacaine in U.S guided TAP block for preemptive analgesia In patients undergoing lower abdominal cancer surgeries.

DETAILED DESCRIPTION:
The transversus abdominis plane (TAP) involves innervations of the anterolateral abdominal wall derived from T6-L1. The block can be given either by anatomical landmark technique or by using an ultrasound probe. The local anesthetic is deposited in a plane between internal oblique and transversus abdominis muscle. It provides adequate postoperative analgesia following various abdominal surgeries.Dexmedetomidine is an alpha-2 agonist that has been approved as a venous sedative and an adjuvant for pain relief .In previous studies, the addition of dexmedetomidine to bupivacaine in the TAP block has prolonged the effect of this block . So far, the optimal dose of dexmedetomidine for the TAP block has not been determined.

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 65 years old
* lower abdominal cancer surgery

Exclusion Criteria:

* patient refusal
* the local anesthetic allergy
* coagulopathy
* local infection at the procedure site
* psychic patients
* patient on chronic opioid use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption during the first 24 hours postoperatively | First 24 hours postoperative
  Morphine consumption during the First 24 hours postoperative

SECONDARY OUTCOMES:
Severity of pain using Visual analogue scale | First 24 hours postoperative
  The severity of pain at rest and on coughing will be assesd using a 10-cm vas(0 means no pain ,10 means worst pain)
Patient level of sedation using four point modified ramsy scale | First 24 hours postoperative
  using a 4-point scale (0 = awake and alert, 1 = minimally sedated, responds to speech, 2 = moderately sedated, arousable by tactile stimulation, and 3 = deeply sedated, arousable only by painful stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Kerolos S Tawfeek, Principal Investigator — Assiut University
Locations (1):
- South egypt cancer institute,Assiut University, Asyut, Egypt